CLINICAL TRIAL: NCT06479018
Title: Identification and Functional Characterization of the Cellular and Molecular Actors of the IL-17B/IL-17RB Axis in Bullous Pemphigoid
Brief Title: Deciphering IL-17-dependant Inflammatory Response in Bullous Pemphigoid
Acronym: BP-IL17RB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PO21096
Record Dates: First submitted 2024-06-14; First posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Bullous Pemphigoid
Keywords: Bullous pemphigoid; IL-17 family; inflammatory response
MeSH Terms: conditions — Pemphigoid, Bullous | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with Bullous Pemphigoid (Experimental)
  Interventions: Biological: Blood sampling; Biological: Liquid bubble sampling; Procedure: Cutaneous biopsy
- Control subjects (Experimental)
  Interventions: Biological: Blood sampling

INTERVENTIONS:
Biological: Blood sampling — Venous blood sampling will be carried out for each patient included in the study.
Biological: Liquid bubble sampling — Liquid bubble sampling will be carried out for each patients with Bullous Pemphigoid included in the study.
  Arms: Patients with Bullous Pemphigoid
Procedure: Cutaneous biopsy — At least the first cutaneous biopsy will be carried out for each patients with Bullous Pemphigoid included in the study.
  Arms: Patients with Bullous Pemphigoid

SUMMARY:
Bullous pemphigoid (BP) is the most frequent autoimmune skin disease and mainly affects elderly individuals. BP classically manifests with tense blisters over urticarial plaques on the trunk and extremities accompanied by intense itches. However, BP is characterized by a large spectrum of clinical presentations allowing to distinguish between typical (with blisters) and atypical forms (non bullous, mucosal damage).

High potency topical steroids and systemic steroids are the current first line intention treatments. While very efficient, these therapies are non-targeted and cause numerous side-effects, especially in these elderly patients that are the most affected. Furthermore, around 30% of BP patients will relapse during the first year of treatment when corticotherapy is decreased or stopped.

The investigators and others have highlighted the presence of Il-17 family belonging-inflammatory cytokines in BP patients. Their functions in the amplification of the inflammatory response and in the mechanisms of relapse have to be precisely determined in order to develop innovative therapeutic approaches and to move forwards precision medicine.

DETAILED DESCRIPTION:
This is a pathophysiological study with prospective and monocentric inclusion.

90 patients with bullous phemphigoid will be recruited from the department of dermatology at the Reims University Hospital.

The main objectives of this study are to identify the cellular and molecular actors of the IL-17B/IL-17RB axis at diagnosis in patients with bullous pemphigoid and to determine their functions in the pathophysiological mechanisms associated with BP at systemic and in situ levels.

The secondary aims of this research are:

1. To confirm IL-17B concentrations in sera at diagnosis as predictive biomarker of BP outcome under local corticotherapy
2. To study the expression kinetics of IL-17B and its receptor IL-17RB in BP patients under treatment
3. To study the implication of IL-17B/IL-17RB axis in BP relapse
4. To establish inflammatory cell composition profile in skin and blood issued from clinical variants of BP as well as from BP patients during the first year of treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients with Bullous Pemphigoid (BP) using the following criteria: clinical features typical of BP with presence of at least three out of four well-established criteria by Vaillant et al.47; subepidermal blister on skin biopsy; and deposits of IgG and/or C3 in a linear pattern along the epidermal basement membrane zone by direct IF.
* patient agreed to participate to the study
* patient affiliated to the French Healthcare System

Exclusion Criteria:

* patient that does not have the ability to give its written informed consent before inclusion in the study
* patient with a pemphigoid gestationis
* patient with a relapse of Bullous Pemphigoid
* patient with Bullous Pemphigoid that already received local superpotent corticotherapy during the last 14 days before inclusion or systemic corticoid treatment during the last 28 days before inclusion
* anemic patient (hemoglobin < 10 g/dL)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-02-10 (Actual); Primary Completion 2025-01-10 (Estimated); Study Completion 2026-01-10 (Estimated)

PRIMARY OUTCOMES:
Identification of IL-17RB-expressing cells and IL-17B-producing cells in blood | Day 1
  Identification of IL-17RB-expressing cells and IL-17B-producing cells in blood from whole blood of patients with BP or control subjects using flow cytometry
Identification of IL-17RB-expressing cells and IL-17B-producing cells in blood | Day 30
  Identification of IL-17RB-expressing cells and IL-17B-producing cells in blood from whole blood of patients with BP or control subjects using flow cytometry
Identification of IL-17RB-expressing cells and IL-17B-producing cells in blood | Day 60
  Identification of IL-17RB-expressing cells and IL-17B-producing cells in blood from whole blood of patients with BP or control subjects using flow cytometry
Identification of IL-17RB-expressing cells and IL-17B-producing cells in blood | Day 90
  Identification of IL-17RB-expressing cells and IL-17B-producing cells in blood from whole blood of patients with BP or control subjects using flow cytometry
Identification of IL-17RB-expressing cells and IL-17B-producing cells in blood | Day 150
  Identification of IL-17RB-expressing cells and IL-17B-producing cells in blood from whole blood of patients with BP or control subjects using flow cytometry
Identification of IL-17RB-expressing cells and IL-17B-producing cells in blood | Day 270
  Identification of IL-17RB-expressing cells and IL-17B-producing cells in blood from whole blood of patients with BP or control subjects using flow cytometry
Identification of IL-17RB-expressing cells and IL-17B-producing cells in blood | Day 365
  Identification of IL-17RB-expressing cells and IL-17B-producing cells in blood from whole blood of patients with BP or control subjects using flow cytometry
Identification of IL-17RB-expressing cells at the lesional site | Day 1
  Identification of IL-17RB-expressing cells at the lesional site from BP skin biopsy specimen harvested using histocytometry
Identification of IL-17RB-expressing cells at the lesional site | Day 60
  Identification of IL-17RB-expressing cells at the lesional site from BP skin biopsy specimen harvested using histocytometry

SECONDARY OUTCOMES:
Measurement of IL-17B concentrations in sera | Day 1
  Measurement of IL-17B concentrations in sera of patients with BP using ELISA technique
Measurement of IL-17B concentrations in sera | Day 30
  Measurement of IL-17B concentrations in sera of patients with BP using ELISA technique
Measurement of IL-17B concentrations in sera | Day 60
  Measurement of IL-17B concentrations in sera of patients with BP using ELISA technique
Measurement of IL-17B concentrations in sera | Day 90
  Measurement of IL-17B concentrations in sera of patients with BP using ELISA technique
Measurement of IL-17B concentrations in sera | Day 150
  Measurement of IL-17B concentrations in sera of patients with BP using ELISA technique
Measurement of IL-17B concentrations in sera | Day 270
  Measurement of IL-17B concentrations in sera of patients with BP using ELISA technique
Measurement of IL-17B concentrations in sera | Day 365
  Measurement of IL-17B concentrations in sera of patients with BP using ELISA technique

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France